CLINICAL TRIAL: NCT06931080
Title: A Phase 2/3, Multicenter, Randomized, Double-blind, Placebo-controlled, Trial to Evaluate the Efficacy and Safety of EB-1020 Once Daily QD XR Capsules Administered Orally at Low or High Dose in Adults With Attention-deficit/Hyperactivity Disorder
Brief Title: Evaluation of the Efficacy and Safety of EB-1020 in Adult ADHD Patients
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 405-102-00112
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 1-(naphthalen-2-yl)-3-azabicyclo(3.1.0)hexane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EB-1020(QD XR capsules) 164.4 mg (Experimental)
  Interventions: Drug: EB-1020 (Centanafadine) 164.4 mg
- EB-1020(QD XR capsules) 328.8 mg (Experimental)
  Interventions: Drug: EB-1020 (Centanafadine) 328.8 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EB-1020 (Centanafadine) 164.4 mg — 164.4 mg, capsule, oral, once daily, for 6 weeks
  Arms: EB-1020(QD XR capsules) 164.4 mg
Drug: EB-1020 (Centanafadine) 328.8 mg — 328.8 mg, capsule, oral, once daily, for 6 weeks
  Arms: EB-1020(QD XR capsules) 328.8 mg
Drug: Placebo — Placebo, capsule, oral, once daily, for 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and examine the safety of two doses of EB-1020 QD XR capsule administered once daily orally in adult ADHD patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed primarily with ADHD (excluding other specified or unspecified attention-deficit/hyperactivity disorder) according to DSM-5 criteria, based on information collected through interviews using the Japanese version of the Conners' Adult ADHD Diagnostic Interview for DSM-IVTM (CAADID).
* Participants with an AISRS total score meeting the following criteria:

  * Not receiving medication treatment for ADHD: 28 points or higher
  * Receiving medication treatment for ADHD: 22 points or higher

Exclusion Criteria:

* Participants who are pregnant or breastfeeding, and those who test positive for pregnancy at screening.
* Participants have a current comorbid psychiatric disorder that either could be expected to require treatment with medications prohibited in this trial, or to confound efficacy or safety assessments. Examples include, but are not limited to, psychotic disorder (current or lifetime), bipolar disorder (current or lifetime), generalized anxiety disorder, obsessive-compulsive disorder, panic disorder, a current major depressive episode, or posttraumatic stress disorder, as established by the MINI.
* Participants diagnosed with a personality disorder according to DSM-5 criteria.
* Participants diagnosed with autism spectrum disorder according to DSM-5 criteria.
* Participants diagnosed with intellectual disability and an IQ score below 70.
* Participants who, in the judgment of the principal or sub-investigator, or based on the following criteria, are at significant risk of suicide:

  • Clear suicidal ideation or a history of suicidal behavior (within the past 6 months) as indicated by a ""yes"" answer to questions 4 or 5 in the suicidal ideation section of the C-SSRS Baseline/Screening version at screening.
* Participants who have a current or past episode of substance-related disorders (excluding tobacco-related disorders) according to DSM-5 diagnostic criteria.
* Participants diagnosed with eating disorders and feeding disorders according to DSM-5 diagnostic criteria.
* Participants who show a positive reaction in alcohol tests or urine drug tests at screening.
* Participants with complications or a history of the following neurological disorders:

  * Epilepsy
  * Seizures (other than infantile febrile seizures)
  * Syncope
  * Tourette's disorder
  * History of significant head trauma with clinically significant loss of consciousness
  * Dementia
  * Cerebrovascular disease
  * Parkinson's disease
  * Intracranial lesions
  * Other severe neurological disorders
* Participants with complications or a history of cardiovascular diseases.
* Participants with clinical laboratory test results at screening that meet any of the following criteria:

  * Platelets <= 75,000/mm3
  * Hemoglobin <= 9 g/dL
  * Neutrophils, absolute <= 1000/mm3
  * AST > 2 x ULN
  * ALT > 2 x ULN
  * Creatinine >= 2 mg/dL
  * CPK >= 2 x ULN (except for the cases that the medical monitor determined that participant's inclusion is possible based on the discussion about the participant's condition with the investigator or subinvestigator) •Abnormal values for both free T4 and TSH•
* Participants who cannot agree to discontinuation of prohibited concomitant medication, such as ADHD medication or antidepressants.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 630 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Adult ADHD Investigator Symptom Rating Scale (AISRS) score at Week6 | Baseline, Weeks 6
  The Adult Investigator Symptom Rating Scale (AISRS) is an 18-item clinician rating scale to evaluate individual ADHD symptoms on a scale of 0 (none) to 3 (severe). The total sum ranges from 0 (no ADHD symptoms) to 54 (extremely severe ADHD symptoms). Negative change from Baseline indicates improvement. Mixed-effect model repeated measure (MMRM) was used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Nobuhito Sanada, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Maynds Tower Mental Clinic, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.